CLINICAL TRIAL: NCT02015377
Title: Food, Adolescence, Mood and Exercise
Brief Title: Food, Adolescence, Mood, and Exercise
Acronym: FAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Donna Spruijt-Metz, Associate Professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: FAME-HS-0700735; 5P60MD002254-04 (NIH)
Record Dates: First submitted 2013-12-09; First posted 2013-12-19 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Sugar/Low Fiber (HSLF) meals (Experimental): Comparing the impact of High sugar/Low fiber (HSLF) meal versus Low Sugar/High Fiber meals (LSHF) on insulin and glucose profiles, gut hormones (ghrelin, amylin, leptin) free fatty acids, cortisol, mood (MOOD), meaning of physical activity (MEANPA), and physical activity engagement (PA) in overweight African American and Hispanic youth
  Interventions: Other: High sugar versus low sugar meals
- Low Sugar/High Fiber (LSHF) meals (Experimental): Comparing the impact of High sugar/Low fiber (HSLF) meal versus Low Sugar/High Fiber meals (LSHF) on insulin and glucose profiles, gut hormones (ghrelin, amylin, leptin) free fatty acids, cortisol, mood (MOOD), meaning of physical activity (MEANPA), and physical activity engagement (PA) in overweight African American and Hispanic youth
  Interventions: Other: High sugar versus low sugar meals

INTERVENTIONS:
Other: High sugar versus low sugar meals — Participants visit our lab for two 8-hour periods with a minimum of two weeks washout in between. In one visit they receive high sugar low fiber meals, in the other they receive low sugar, high fiber meals. The order of meals is randomized

SUMMARY:
The overall objective of FAME is to examine the metabolic and behavioral links between dietary intake and its subsequent effects on circulating appetite regulating hormones and physical activity levels in Hispanic and African American adolescents.

DETAILED DESCRIPTION:
Our major unifying hypothesis is that diets comprised of high sugar, energy dense, low fiber meals, are associated with a post-prandial metabolic, hormonal and psychosocial profile that promotes overeating and sedentary behavior. Specific Aims: (1) Compare the effects of a HIGH SUGAR, LOW FIBER (HSLF) meal versus a LOW SUGAR, HIGH FIBER (LSHF) meal on insulin dynamics, selected gut peptides, mood and levels of physical activity in minority adolescents, (2) Explore the effects of HSLF versus LSHF meals on post-prandial ad libitum food intake, (3) Explore differences in reaction to HSLF versus LSHF meals in lean and overweight adolescents and (4) Examine ethnic differences in meal responses between Hispanic and African American children. Research Design and Methods: We will employ a cross-over design with a 3-4 week washout period where normal weight and overweight African American and Hispanic youth come to our Observation Lab in a fasting state and consume high sugar and low sugar meals at separate visits in random order. Meal consumption will be followed by five hours of intensive observation in which we quantify real-time physical activity in laboratory setting that was designed to offer equally attractive choices for active or sedentary behaviors. After 5 hours, participants will be offered food platters with an array of food types and be invited to eat ad libitum. Subsequent energy and nutrient intake will be quantified. Rationale: This study is prompted by three observations: (1) The disproportionate levels of obesity and risk for type 2 diabetes and cardiovascular disease in Hispanic and African American children; (2) The rapid decline in physical activity during puberty especially in Hispanic and African American adolescents, and (3) Children, and particularly minority children, tend to have diets high in added sugars and low in fiber. Thus, it is imperative to improve our understanding of the interrelationships between dietary intake, physical activity and risk factors for type 2 diabetes and cardiovascular disease in minority youth, particularly during puberty, when physical activity levels significantly decline. Relevance to public health: This study will provide new information on the acute effects of meal composition on mood and subsequent choices of physical activity in normal weight, healthy overweight and insulin resistant overweight Hispanic and African American youth. Furthermore, we suggest that our findings may potentially lead to a better understanding the acute affects of poor nutritional choices on physical activity in minority adolescent populations at high risk for obesity, diabetes type 2, and other obesity-related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Children (9th - 11th grade, ~14-17yrs)
* Male and female
* Hispanic or African American

Exclusion Criteria:

* Diabetes
* Currently in weight loss or exercise program
* BMI < 85th percentile as defined by CDC growth curves
* Use of medications that influence body weight or SI
* Syndromes that influence body composition

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2007-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
changes in physical activity as measured by accelerometer over an 8 hour in lab visit | physical activity is measured continuously by accelerometer worn on belt
  Physical activity is measured by an actigraph accelerometer which is worn over the right hip on a belt.

SECONDARY OUTCOMES:
Changes in blood glucose levels over 5 hours | Every 30 minutes for 5 hours
  On the day of the meal visits, participants arrived at the Observation Lab on campus at approximately 7:00 am after a 10-hour overnight fast. Topical anesthetic (EMLA) will immediately be placed on likely forearm IV sites. After every effort has been made to "break the ice" and develop rapport, a saline lock intravenous catheter was inserted and secured for stability in a forearm vein, not involving wrist or elbow joint in order to maximize motility during free activity. After a baseline blood draw (at -5 min), participants will be provided with a breakfast test meal. Blood is drawn every 30 minutes for 5 hours. The saline lock and blood draws were conducted by a trained and certified nurse.
Changes in insulin over 5 hours | Blood was drawn every 30 minutes for 5 hours
  On the day of the meal visits, participants arrived at the Observation Lab on campus at approximately 7:00 am after a 10-hour overnight fast. Topical anesthetic (EMLA) will immediately be placed on likely forearm IV sites. After every effort has been made to "break the ice" and develop rapport, a saline lock intravenous catheter was inserted and secured for stability in a forearm vein, not involving wrist or elbow joint in order to maximize motility during free activity. After a baseline blood draw (at -5 min), participants will be provided with a breakfast test meal. Blood is drawn every 30 minutes for 5 hours. The saline lock and blood draws were conducted by a trained and certified nurse.
Stress (objective and perceived) fluctuations over 5 hours | Every 30 minutes for 5 hours
  Every 30 minutes at the time of the blood draws, salivary cortisol was measured by salivette and perceived stress was measured by validated Visual Analogue Scale

CONTACTS AND LOCATIONS:
Overall Officials: Donna Spruijt-Metz, Ph.D, Principal Investigator — University of Southern California; Michael I Goran, Ph.D, Study Director — University of Southern California
Locations (1):
- University of Southern California Health Science Campus, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided